CLINICAL TRIAL: NCT05392387
Title: Study on the Antiviral Therapy and Prognosis of Patients With Chronic HBV Infection
Brief Title: Treatment and Prognosis of Patients With Chronic HBV Infection
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yan Huang, MD, Professor, Xiangya Hospital of Central South University
Other Study IDs: Xiangya HBV project
Record Dates: First submitted 2022-05-17; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B Virus Infection
Keywords: Hepatitis B Virus Infection; antiviral therapy; prognosis
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood including blood cells, serum and plasma, urine, faeces and liver tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- peg-IFN-alpha alone: Patients with chronic HBV infection only treated with peg-IFN-alpha
  Interventions: Other: Standard antiviral therapy
- nucleos(t)ide analogues alone: Patients with chronic HBV infection only treated with nucleos(t)ide analogues
  Interventions: Other: Standard antiviral therapy
- combination: Patients with chronic HBV infection treated with nucleos(t)ide analogues and peg-IFN-alpha
  Interventions: Other: Standard antiviral therapy

INTERVENTIONS:
Other: Standard antiviral therapy — pegylated interferon or/and nucleos(t)ide analogues

SUMMARY:
Hepatitis B virus (HBV) infection is a major global health issue with 257 million chronically infected individuals. Of note, China has the largest population accounting for one third of the world's infected population. Approximately, about 300 000 people die each year due to the consequences of HBV. In 2016, the World Health Organization (WHO) proposed the goal for elimination of hepatitis B as public health threat by 2030 and China will be a major contributor towards this global goal. Currently, two approved therapeutic strategies are available including pegylated interferon (IFN) or nucleos (t) ide analogues (NA), which could suppress HBV replication and slow disease progression. Here, investigators hope to launch a cohort study to reveal the clinical features relating to therapeutic efficacy of antiviral therapy and the prognosis of patients with differential therapeutic strategies.

DETAILED DESCRIPTION:
Patients with chronic HBV infection were recruited in the current study and divided in to peg-IFN-alpha alone group, NAs alone group and the combination therapy group. The serum HBV DNA level, HBV serological test and biochemical examination including serum transaminase level and AFP were recorded every three or six months. The serum, feces, urine and liver (if necessary) samples were collected during follow-up. And the clinical outcomes of patients were evaluated. The clinical and biological features of patients with different clinical outcomes will be compared to explore the factors affecting the antiviral therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

patients with evidence of chronic HBV infection

Exclusion Criteria:

chronic liver injury mainly caused by other reasons, such as autoimmune diseases, alcohol, drugs and so on.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The chronic HBV-infected patients with differential antiviral strategies were recruited and separated to peg-IFN-alpha alone, NAs alone or combination treatment groups according to their antiviral therapies. The clinical outcomes of patients with differential treatments were compared during the follow-up management.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
virological response | 3 years
  serum HBV DNA level below the detection limit
HBeAg seroconversion | 3 years
  Loss of HBeAg and presence of anti-hepatitis B e antibody (anti-HBe) in a person who was previously HBeAg-positive and anti-HBe-negative
Clinical cure | 3 years
  Sustained virological response and HBsAg clearance or with anti-HBs seroconversion, alanine aminotransferase (ALT) within the normal range, and mild or no lesions in the liver

SECONDARY OUTCOMES:
HBV DNA | 3 years
  The serum HBV DNA level will be detected and reported every 3 to 6 months
HBV serological test | 3 years
  HBV serological markers include HBsAg, anti-HBs, HBeAg, anti-HBe, hepatitis B core antibody (anti-HBc) were detected and reported every 3 months
liver function | 3 years
  The serum levels of transaminase including ALT and aspartate aminotransferase (AST) will be collected and reported every 3 months
Alpha-fetoprotein (AFP) | 3 years
  The serum AFP level will be detected and reported every 3 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Huang, Study Director — Xiangya Hospital of Central South University
Locations (1):
- Department of Infectious Disease, Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided